CLINICAL TRIAL: NCT01972347
Title: An Open Label, Single Centre, Phase II Pilot Study of Neoadjuvant Dabrafenib + Trametinib in Patients With Resectable American Joint Committee on Cancer (AJCC) Stage IIIB-C BRAF V600 Mutation Positive Melanoma
Brief Title: Neoadjuvant Dabrafenib + Trametinib for AJCC Stage IIIB-C BRAF V600 Mutation Positive Melanoma
Acronym: Neo Combi
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Melanoma Institute Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200332
Record Dates: First submitted 2013-06-17; First posted 2013-10-30 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Melanoma
Keywords: Melanoma; Cutaneous melanoma; Malignant melanoma; Stage III B / C melanoma; Neoadjuvant treatment; Pyrexia; Biomarkers; Dabrafenib; Trametinib
MeSH Terms: conditions — Melanoma; Fever | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dabrafenib and Trametinib (Experimental): Dabrafenib 150mg bid orally and Trametinib 2mg od orally for 52 weeks
  Interventions: Drug: Dabrafenib; Drug: Trametinib

INTERVENTIONS:
Drug: Dabrafenib — Patients will receive neoadjuvant treatment with dabrafenib 150mg twice a day and trametinib 2mg once a day for 12 weeks. Patients will then have complete lymph node dissection and will continue on maintenance treatment with dabrafenib 150mg twice a day and trametinib 2mg once a day for 40 weeks.
  Other Names: GSK2118436
Drug: Trametinib — Patients will receive neoadjuvant treatment with dabrafenib 150mg twice a day and trametinib 2mg once a day for 12 weeks. Patients will then have complete lymph node dissection and will continue on maintainance treatment with dabrafenib 150mg twice a day and trametinib 2mg once a day for 40 weeks.
  Other Names: GSK1120212

SUMMARY:
This is an open label, single centre, phase II study of neoadjuvant drug treatment with dabrafenib + trametinib in patients with resectable American Joint Committee on Cancer (AJCC) Stage IIIB-C BRAF V600 mutation positive melanoma.

The main aim of this study is to find out if giving of a new combined drug treatment to patients with melanoma that has spread to the lymph nodes BEFORE they have surgery, will result in improved clinical and pathological response of the melanoma tissue after 12 weeks treatment.

DETAILED DESCRIPTION:
Neoadjuvant therapy has been demonstrated to improve outcome in the management of patients of multiple different solid tumours. The advantage of a neoadjuvant therapy in melanoma is that it provides in vivo assessment of tumour responsiveness to systemic therapy, potentially eradicates micrometastatic disease, and may improve the surgical result. It also provides an opportunity to obtain tumour samples before and after treatment to study variation of response and effects of treatment on tumour characteristics.

This pilot study explores pathological response rates, Response Evaluation Criteria in Solid Tumors (RECIST) response rates and biomarkers for a 12-week duration of neoadjuvant therapy with combined MAP kinase inhibition (MAPKi) with dabrafenib and trametinib and to establish guidelines for an expanded Phase II or III study.

The biomarker component of this study will compare pre-treatment (PRE) with day 4-7, 'early during treatment' biopsies (EDT) and 12 week lymphadenectomy samples (POST). The tissue will be interrogated for immunologic, proteomic and genetic (RNA and DNA) features and changes in tissue and blood. The baseline PRE specimen will consist of at least two core, excisional or incisional biopsies taken prior to commencing combined dabrafenib and trametinib. The EDT specimen will consist of at least two core, excisional or incisional biopsies taken at days 4-7, very early after commencing combined dabrafenib and trametinib. The POST specimen will be the complete lymph node dissection specimen performed after 12 weeks of treatment with combined dabrafenib and trametinib.

The EDT specimen provides a unique opportunity to investigate the early changes that occur in a melanoma tumour with MAPK inhibitors that may set up for later resistance or complete response, and that may be amenable to therapeutic manipulation. For example, EDT samples collected on patients treated with single agent BRAF inhibitors showed increased T cell infiltrate that was associated with a better response in the lesion. The T cell infiltrate has also been associated with increased expression of melanoma antigens, a decrease in immunosuppressive cytokines [interleukin (IL)-6 and IL-8] and an increase in markers of T-cell cytotoxicity. Additional studies have shown the expected suppression in pERK, and in paired PRE-EDT samples, the decreased ERK suppression is associated with a better RECIST response. There have been no reports of the effects of BRAF and MEK inhibitors as single agent or in combination on responding melanoma tissue taken more than 15 days after commencement of treatment. As the median PFS for the combination of dabrafenib and trametinib is 9.4 months, >95% of the POST samples will be responding, and provide an opportunity to 1) compare the responding POST with the EDT sample (and the baseline PRE samples prior to treatment) to investigate how signalling pathways (as determined by RNA gene expression and protein expression) alter with time, and 2) how the changes in signalling pathways correlate with clinical and pathological response.

Study treatment will be continued as adjuvant therapy. The goal is to improve the cure rate after surgery through eradication of occult micrometastatic disease. Notable successes have been achieved in oncology when highly effective therapies were available for advanced stage disease (e.g., breast cancer, Hodgkin's and non-Hodgkin's lymphoma, embryonal tumours, osteosarcoma). High-risk, resected BRAF V600 mutation positive melanoma represents another attractive setting for testing this paradigm since: 1) the population is at high risk for relapse and death without further therapy and 2) the BRAF/MAP-ERK kinase combination is highly effective in the metastatic setting and can be targeted to the population most likely to benefit. The study design will test the efficacy of study treatment in both the neoadjuvant and adjuvant settings for the first time in this patient population.

Approximately 168 patients have received combination therapy with dabrafenib and trametinib at the proposed study doses (150 mg BID dabrafenib and 2 mg once daily trametinib) with a median follow-up time of 12.8 months. In the dose-escalation phase, PFS was longest for the group receiving the highest doses of dabrafenib and trametinib with an acceptable safety profile. Based on these data the combination of 150 mg BID of dabrafenib and 2.0 mg once daily of trametinib has been selected for this study. Mature randomized phase 2 trial (Part C in Figure 2 above) with a median follow up of 14.1 months showed a higher response rate (76% versus 54%, p=0.03) and a longer median PFS (9.4 months vs 5.8 months, hazard ratio (HR) 0.39, p<0.001) in MAPK inhibitor-naïve patients on the combination of the full dose of dabrafenib and trametinib compared with dabrafenib monotherapy.

The duration of therapy (12 months) is based upon expert consensus and does not exceed that administered in other pivotal studies of adjuvant treatment in similar populations where treatment ranged from 12 to 60 months. In the absence of a reliable biomarker for minimal residual disease, empiric dosing for durations much shorter than the predicted median relapse free interval (median of 15 months) may increase the risk of treatment failure. The design does include predictive biomarkers which may allow further refinement of dosing once a phase III study of this design has been completed. Safety of continuous dosing of dabrafenib and trametinib for over a year as monotherapies has been established along with preliminary safety of combination dosing for a similar interval. Safety precautions will include clear guidelines for management of toxicity, including enhanced surveillance for adverse events of special interest along with instructions for dose modification. The inclusion/exclusion criteria will also serve to minimize participation of those at greatest risk for known or suspected toxicities of the combination therapy.

Neoadjuvant studies in patients with macroscopic stage III melanoma have been performed using the immunotherapies interferon and ipilimumab. Interferon has no activity in stage IV melanoma, yet there was an objective clinical response in 11 of 17 (55%) patients with stage III melanoma when given neoadjuvantly. Furthermore, 3/17 (15%) had a complete pathological response. Clinical responders had significantly greater increases in endotumoral CD11c and CD3 cells and significantly greater decreases in endotumoral CD83 cells compared with nonresponders. In contrast, ipilimumab confers an overall survival benefit for patients with stage IV melanoma over vaccine or chemotherapy, however the objective response rate is low at 11-15%. In the neoadjuvant study with macroscopic stage III melanoma, pathological responses were not reported, however objective clinical responses were observed in 3/29 (10%) patients. Immune infiltrate cells were noted in most tumours after treatment with ipilimumab, and results correlating biomarker changes with response are awaited.

In stage IV melanoma patients, over 73% of patients who respond to BRAF inhibitors, will achieve a RECIST response by the time of the first scan (8 weeks), and the median time to best response is 12 weeks in the poorest prognosis patients. The progression free survival (PFS) for the combination is 9.4 months, and <5% of patients have progression as their best RECIST response. Therefore, 12 weeks was chosen for the period of neoadjuvant combination therapy to optimise tumour shrinkage, without compromising patient safety.

Surgeons at the Melanoma Institute Australia perform approximately 120 lymphadenectomies each year for patients with palpable lymphadenopathy. The sample size of 35 patients is achievable within the anticipated 12 to 18 month recruitment phase. Neoadjuvant therapy with combined dabrafenib + trametinib for these high-risk melanoma patients with bulky regional stage IIIB-C lymphadenopathy may result in improved rates and duration of local control with reduced surgical morbidity.

Pyrexia Sub-Study Combined therapy with dabrafenib and trametinib is associated with pyrexia in over two-thirds of patients. There are no identifiable clinical correlates of pyrexia and the mechanism remains unknown. Management involves the use of corticosteroids in 25% of cases. Further investigations of this drug-associated pyrexia are urgently required, particularly for facilitating the use of these drugs in the adjuvant setting. The context of this single institution study with its close and uniform patient monitoring provides an ideal opportunity to study drug-induced pyrexia, its mechanisms, prevention and management, and correlation of pyrexia with parent drug and metabolite plasma levels compared with those who do not develop pyrexia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically confirmed AJCC Stage IIIB or IIIC (Tx, T1-4, N1b, N2b, N2c, N3, Mo) cutaneous melanoma or unknown primary determined to be BRAF V600 mutation positive, with sufficient nodal or in-transit disease to enable biopsies prior to surgery.Patients must have disease that is measurable per RECIST version 1.1
* Able to swallow and retain oral medication and must not have any clinically significant gastrointestinal abnormalities that may alter absorption
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Adequate baseline organ function
* Women of childbearing potential must have a negative serum pregnancy test within 7 days of first dose of study treatment and agree to use effective contraception from 14 days prior to commencing study treatment, throughout the treatment period and for 4 months after the last dose of study treatment
* Men with any female partner of childbearing potential must agree to use effective contraception from 14 days prior to commencing study treatment, throughout the treatment period and for 4 months after the last dose of study treatment

Exclusion Criteria:

* Known mucosal or ocular melanoma or any unresectable in-transit metastases
* Evidence of distant metastatic disease on screening evaluation
* Prior anti-cancer treatment for melanoma (chemotherapy, immunotherapy, biologic therapy, vaccine therapy, investigational treatment or radiotherapy). Prior surgery for melanoma is allowed.
* Taken an investigational drug within 28 days or 5 half-lives, whichever is longer, prior to commencing study treatment.
* Current or expected use of a prohibited medication(s)
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study treatments, their excipients, and/or dimethyl sulfoxide (DMSO)
* Known HIV
* A history of known glucose-6-phosphate dehydrogenase (G6PD) deficiency
* History of another malignancy or a concurrent malignancy except:

  1. Patients who have been disease-free for 3 years and have a life expectancy of > 5 years;
  2. Patients with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible, for example cervical cancer in situ, atypical melanocytic hyperplasia or melanoma in situ, multiple primary melanomas.
* A history or evidence of cardiovascular risk including any of the following: a. QT interval corrected for heart rate using the Bazett's formula ≥480 msec or ≥ 450 msec for patients with bundle branch block; b. History or evidence of current clinically significant uncontrolled arrhythmias; c. History of acute coronary syndromes (including myocardial infarction or unstable angina), coronary angioplasty, or stenting within 6 months prior to commencement of study treatment; d. History or evidence of current ≥ Class II congestive heart failure; e. Abnormal cardiac valve morphology documented by echocardiogram which in the opinion of the investigator could interfere with the patient's safety.

  f. Treatment refractory hypertension defined as a blood pressure of systolic > 140 mm Hg and/or diastolic > 90 mm Hg which cannot be controlled by anti-hypertensive therapy.
* A history or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR)
* Any serious or unstable pre-existing medical conditions (aside from the malignancy exceptions specified above), psychiatric disorders, or other conditions that, in the opinion of the treating clinician, could interfere with the patient's safety, obtaining informed consent, or compliance with study procedures.
* Breastfeeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of viable melanoma tissue, compared to baseline, in dissected lymph node and / or in-transit tumour tissue after 12 weeks of neoadjuvant treatment. | 12 weeks
  The proportion of viable melanoma tissue, compared to baseline, in dissected lymph node and / or in-transit tumour tissue after 12 weeks of neoadjuvant treatment.

SECONDARY OUTCOMES:
Effects of neoadjuvant study treatment on surgical outcomes after complete lymph node and / or in-transit disease dissection. | 12 weeks
  Number of episodes (and patient number) of infection at wound site requiring intravenous antibiotics and wound drainage, duration of time from surgery to removal of drain because of ceased or minimal drainage, number of episodes (and patient number) of seroma formation at wound site requiring any intervention and volume of seroma drainage, number of episodes (and patient number) of bleeding .from wound requiring return to theatre or transfusion(s), bioimpedance measures of limb distal to site of CLND (axilla and groin only) at baseline, and weeks 8, 24 and 40 after CLND (20, 40 and 52 weeks after starting study treatment) and correlation of surgical outcomes with response to study treatment.
Effects of study treatment on host immune response in tumour tissue and peripheral blood. | 12 weeks
  Immune tumour tissue will be assessed as outlined in 3b and 3c. Peripheral blood will be examined for levels of cytokines and chemokines (Millipore multiplex) and changes in host immune response in tumour and peripheral blood will be correlated with pathological and clinical response.
Correlation of pyrexia episodes and signs with baseline melanoma disease burden (number and size of lymph nodes), RECIST response, pathological response, immune related changes in tumour tissue and peripheral blood. | 52 weeks
  Correlation of pyrexia episodes and signs with baseline melanoma disease burden (number and size of lymph nodes), RECIST response, pathological response, immune related changes in tumour tissue and peripheral blood.
Description of specific blood and serum changes that occur with pyrexia. | 52 weeks
  Measurement of the following, at regular intervals in all patients, with or without pyrexia, and at every febrile episode: serum chemokines and cytokines, including IL-1, IL6, IL-8, IL-10, IL-18, PD1, gamma interferon and TNF-alpha; plasma and serum parent and metabolite concentrations, white blood cell subsets, liver function tests; AST, ALT, Bilirubin, full blood count, other changes such as cortisol, adrenocorticotropic hormone.
Relapse free survival | 52 weeks plus the time when 70% of patients have died
  Relapse free survival defined as the interval from commencement of study treatment to local or distant recurrence with censoring of patients dying from causes other than melanoma or treatment related toxicity at date of death. Patients alive without recurrence or with second primary cancers will be censored at date of last assessment. A second primary melanoma will not be considered relapse.
Overall survival | 52 weeks plus until the time that 70% of patients have died
  Overall survival defined as the interval from commencement of study treatment to the date of death. Patients still alive will be censored at the date of last follow up (until 70% of patients have died)
Description of adverse events and how these correlate with clinical outcomes | 52 weeks
  Description of adverse events and how these correlate with clinical outcomes
The clinical response to 12 weeks neoadjuvant treatment | 12 weeks
  The clinical response will be measured according to the Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1
Correlation of a range of tumour biomarkers at baseline, early treatment and 12 week intervals with pathological and clinical response. | 12 weeks
  Immunohistochemistry; including, but not restricted to CD3, CD4, CD8, FOXP3, PD-L1, PD-1, Tunel assay (apoptosis), macrophages (CD68, CD163), Ki67, cyclin D1, pERK, p27, p21, p16, SROUTY, DUSP 4and6, pAKT, MITF, beta-catenin, PDGFR, EGFR, IGFR, MCL-1, BCL-2, p53, Gramzyme B, CD20, CD1a. RNA expression profile baseline (PRE), early treatment (EDT) and at 12 weeks POST), DNA mutation analysis, DNA copy number analysis, DNA methylation pattern, PRE and/or POST, DNA methylation pattern and proteomic profiling in PRE and POST samples.

CONTACTS AND LOCATIONS:
Overall Officials: Georgina Long, Study Director — Melanoma Institute Australia
Locations (1):
- Melanoma Institute Australia, Wollstonecraft, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No
If approached, we would be happy to consider making IPD available.

REFERENCES:
- [Derived] Long GV, Saw RPM, Lo S, Nieweg OE, Shannon KF, Gonzalez M, Guminski A, Lee JH, Lee H, Ferguson PM, Rawson RV, Wilmott JS, Thompson JF, Kefford RF, Ch'ng S, Stretch JR, Emmett L, Kapoor R, Rizos H, Spillane AJ, Scolyer RA, Menzies AM. Neoadjuvant dabrafenib combined with trametinib for resectable, stage IIIB-C, BRAFV600 mutation-positive melanoma (NeoCombi): a single-arm, open-label, single-centre, phase 2 trial. Lancet Oncol. 2019 Jul;20(7):961-971. doi: 10.1016/S1470-2045(19)30331-6. Epub 2019 Jun 3. PMID 31171444
- [Derived] Kim HY, Duong JK, Gonzalez M, Long GV, Menzies AM, Rizos H, Lim SY, Lee J, Boddy AV. Pharmacokinetic and cytokine profiles of melanoma patients with dabrafenib and trametinib-induced pyrexia. Cancer Chemother Pharmacol. 2019 Apr;83(4):693-704. doi: 10.1007/s00280-019-03780-y. Epub 2019 Jan 19. PMID 30661097
- See also: Melanoma Institute Australia - current research projects — http://www.melanoma.org.au/research/current-projects/